CLINICAL TRIAL: NCT05784987
Title: An Open, Single-arm, Multi-center Clinical Trial of Molecular Subtype-guided R-MINE+X Regimen in the Treatment of Relapsed/Refractory Diffuse Large B-cell Lymphoma (DLBCL)
Brief Title: R-MINE+X in Patients With Relapsed/Refractory Diffuse Large B-cell Lymphoma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSPC-DED-DLBCL-K09
Record Dates: First submitted 2023-03-02; First posted 2023-03-27 (Actual); Last update posted 2023-03-27 (Actual); Status verified 2023-03

CONDITIONS: Diffuse Large B-cell Lymphoma
Keywords: DLBCL; R-MINE+X; Mitoxantrone liposome
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — Rituximab; Ifosfamide; Etoposide

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- R-MINE+X (Experimental): R-MINE: Rituximab, Isophosphamide, Mitoxantrone hydrochloride liposome, Etoposide
  X: Orelabrutinib, Chidamide, Penpulimab, Lenalidomide
  Interventions: Drug: Rituximab; Drug: Mitoxantrone hydrochloride liposome; Drug: Isophosphamide; Drug: Etoposide; Drug: X: Orelabrutinib; Drug: X: Chidamide; Drug: X: Penpulimab; Drug: X: Lenalidomide

INTERVENTIONS:
Drug: Rituximab — 375 mg/m2, d0, Cycle 1~4
Drug: Mitoxantrone hydrochloride liposome — 20 mg/m2, d1, Cycle 1~4
Drug: Isophosphamide — 1.33 g/m2, d1-3(Rescue with equal dose of mesperidine), Cycle 1~4
Drug: Etoposide — 65 mg/m2, d1-3, Cycle 1~4
Drug: X: Orelabrutinib — MCD/BN2 subtype: BTK inhibitor-Orelabrutinib: 150 mg/d, d1-21, Cycle 2~4
Drug: X: Chidamide — EZB subtype: Chidamide: 20 mg/d, d1, d4, d8, d11, Cycle 2~4
Drug: X: Penpulimab — TP53 mutation - X: PD-1 monoclonal antibody - Penpulimab: 200mg/d, d0, Cycle 2~4
Drug: X: Lenalidomide — Other-X: Lenalidomide: 25mg/d, d1-10, Cycle 2~4

SUMMARY:
Based on the modified R-MINE of mitoxantrone hydrochloride liposome, the corresponding targeted drug (X) was added according to the genotyping detected by second-generation gene sequencing (NGS) to explore the effectiveness and safety of R-MINE+X in the treatment of recurrent/refractory (R/R) diffuse large B-cell lymphoma (DLBCL).

DETAILED DESCRIPTION:
Compared with traditional mitoxantrone, mitoxantrone liposomes can significantly prolong the survival time of patients and reduce the cardiotoxicity and non-hematological toxicity of anthracycline drugs. At present, there are no studies on the efficacy and safety of R-MINE+X regimen based on molecular typing in the treatment of R/R DLBCL. Therefore, based on NGS, R/R DLBCL was divided into different molecular types (MCD subtype, BN2 subtype, EZB subtype, A53 subtype and other subtype), and on this basis, different molecular types of targeted drugs (X: MCD/BN2 subtype - BTK inhibitor, EZB subtype - Chidamide, A53 subtype - PD-1 monoclonal antibody and other type - lenalidomide) were used to treat R/R DLBCL. The main purpose was to observe the effectiveness and safety of the program in R/R DLBCL.

ELIGIBILITY:
Inclusion Criteria:

1. Join the study voluntarily and sign the informed consent;
2. Age ≤ 18 years old ≤75 years old;
3. Expected survival time ≥3 months;
4. Recurrent or refractory diffuse large B-cell lymphoma confirmed by histopathology;
5. Consistent with relapsed or refractory lymphoma: Relapsed lymphoma refers to lymphoma that relapsed after CR obtained from initial chemotherapy. Refractory lymphoma is diagnosed by meeting any of the following criteria: 1) tumor shrinkage < 50% or progression after 4 courses of chemotherapy prescribed by the standard regimen; 2) CR was achieved by standard chemotherapy, but recurrent within half a year; 3) Relapse for two or more times after CR; 4) Recurrence after hematopoietic stem cell transplantation;
6. There must be at least one evaluable or measurable lesion in line with Lugano2014 criteria: lymph node lesion, the length and diameter of detectable lymph node must be greater than 1.5cm; For non-lymph node lesions, the diameter of extrinsic lesions should be > 1.0cm;
7. ECOG score 0-2;
8. Bone marrow function: neutrophil count ≥1.5×10^9/L, platelet count ≥75×10^9/L, hemoglobin ≥80g/L (neutrophil count ≥1.0×10^9/L, platelet count ≥50×10^9/L, hemoglobin ≥75g/L in patients with bone marrow involvement);
9. Liver and kidney function: serum creatinine ≤1.5 times the upper limit of normal value; AST and ALT ≤2.5 times the upper limit of normal value (≤5 times the upper limit of normal value for patients with liver invasion); Total bilirubin ≤1.5 times the upper limit of normal value (≤3 times the upper limit of normal value for patients with liver invasion);

Exclusion Criteria:

1. The subject's previous history of antitumor therapy meets one of the following conditions:

   1. Previous recipients of mitoxantrone or mitoxantrone liposomes;
   2. Prior treatment with doxorubicin or anthracycline with a cumulative dose of doxorubicin > 360 mg/m2 (1 mg of doxorubicin for other anthracyclines);
   3. Patients who had received autologous hematopoietic stem cell transplantation or had received allogeneic hematopoietic stem cell transplantation within 100 days of the first medication;
   4. Received anti-tumor therapy (including chemotherapy, targeted therapy, hormone therapy, taking anti-tumor active Chinese medicine, etc.) or participated in other clinical trials and received clinical trial drugs within 4 weeks before the first use of the drug in this study;
2. Hypersensitivity to any investigational drug or its components;
3. Uncontrolled systemic diseases (such as advanced infections, uncontrolled hypertension, diabetes, etc.);
4. Cardiac function and disease conform to one of the following conditions:

   1. Long QTc syndrome or QTc interval >480 ms;
   2. Complete left bundle branch block, complete right bundle branch block with left anterior branch block, second degree type II, or third degree atrioventricular block;
   3. severe, uncontrolled arrhythmias requiring medical treatment;
   4. New York College of Cardiology Grade ≥ III;
   5. A history of acute myocardial infarction, unstable angina pectoris, severely unstable ventricular arrhythmias or any other arrhythmia requiring treatment, a history of clinically severe pericardial disease, or electrocardiographic evidence of acute ischemic or active conduction abnormalities within the 6 months prior to recruitment.
5. Hepatitis B and hepatitis C active infection (hepatitis B virus surface antigen positive and hepatitis B virus DNA more than 1x10^3 copies /mL; HCV RNA over 1x10^3 copies /mL);
6. Human immunodeficiency virus (HIV) infection (HIV antibody positive);
7. Past or present co-existing malignancies (in addition to non-melanoma basal cell carcinoma of the skin, carcinoma in situ of the breast/cervix, and other malignancies that have been effectively controlled without treatment in the past five years);
8. Primary or secondary central nervous system (CNS) lymphoma or history of CNS lymphoma at the time of recruitment;
9. There is significant gastrointestinal disease at the time of screening that may affect drug intake, transport or absorption (e.g. inability to swallow, chronic diarrhea, intestinal obstruction, etc.);
10. Pregnant and lactating women and patients of childbearing age who do not wish to take contraceptive measures;
11. Situations in which other researchers have determined that participation in this study is not appropriate.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-04-15 (Estimated); Primary Completion 2024-01-01 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate(ORR) | up to 4 cycles of chemotherapy(each cycle is 21 days)
  Objective response rate (ORR) after 4 cycles of R-MINE+X chemotherapy

SECONDARY OUTCOMES:
Complete remission rate(CRR) | up to 4 cycles of chemotherapy(each cycle is 21 days)
  Complete remission rate(CRR) after 4 cycles of R-MINE+X chemotherapy
Duration of remission(DOR) | up to 4 cycles of chemotherapy(each cycle is 21 days)
  Time from reaching CR or PR for the first time to disease progression
Progression-Free-Survival rate | 1 year
  from date of inclusion to date of progression, relapse, or death from any cause
Overall survival rate | 1 year
  from the date of inclusion to date of death, irrespective of cause
Adverse events (AE) | From the first day of medication to 28 days after the last dose
  The safety of the drug was evaluated by NCI-CTC AE 5.0 standard

CONTACTS AND LOCATIONS:
Overall Officials: Wei Xu, PhD& MD, Principal Investigator — The first Affiliated Hospital Of Nanjing Medical University(JiangSu Province Hospital)